CLINICAL TRIAL: NCT02814864
Title: Clinical Phase II Trial Evaluating the Efficacy of Systemic Mesenchymal Stromal Cell (MSC) Injections for the Treatment of Severe and Chronic Radiotherapy-induced Abdomino-pelvic Complications (Pelvic Radiation Disease, PRD) Refractory to Standard Therapy
Brief Title: Trial Evaluating the Efficacy of Systemic Mesenchymal Stromal Cell (MSC) Injections for the Treatment of Severe and Chronic Radiotherapy-induced Abdomino-pelvic Complications (Pelvic Radiation Disease, PRD) Refractory to Standard Therapy
Acronym: PRISME
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P130935; 2014-001462-99 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-28 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Pelvic Radiation Therapy; Radiation-induced Hemorrhagic Cystitis
Keywords: Hematology; Mesenchymal Stromal Cell; radiotherapy; gastro-intestinal complications; lower digestive tract cancers; colitis; bleeding; diarrhea; pelvic radiation disease
MeSH Terms: conditions — Colitis; Hemorrhage; Diarrhea | interventions — Injections; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stromal Cell (MSC) (Experimental): Patient with chronic radiotherapy-induced abdomino-pelvic complications refractory to standard therapy: 12 patients suffering of PRD (LENT-SOMA scale>2)
  Interventions: Drug: Mesenchymal Stromal Cell (MSC) injections

INTERVENTIONS:
Drug: Mesenchymal Stromal Cell (MSC) injections — 12 patients suffering of PRD (LENT-SOMA scale>2) will receive Mesenchymal Stromal Cell (MSC) injections
  Other Names: Cell therapy

SUMMARY:
Patients receiving radiation therapy are still at risk for side effects due to off-target radiation damage of normal tissues The number of cancer patients is expected to increase from 14.1 million around the world in 2012 to 19.3 million in 2025. Up to ten percent will develop late severe gastrointestinal complications (i.e. Pelvic Radiation Disease - PRD). Symptoms are proctopathy (5-20%) and radiation-induced cystitis (3,5%) that affect quality of life. The treatment of PRD is limited to managing the symptoms; new alternatives should be proposed.

Clinical trials using MSCs to treat hemorrhagic cystitis, proctopathy have demonstrated the feasibility to used MSCs in these pathologies :

* MSCs successfully repair hemorrhagic cystitis, and perforated colon in patients with hemorrhagic cystitis, perforated colon and peritonitis.
* Six clinical trials are currently ongoing for proctopathy, 3 are phase III. Results suggest an inhibition of chronic inflammation and fistulization and interruption of hemorrhagic syndromes.
* Clinical trials to evaluate the efficacy of MSCs to treat hemorrhagic cystitis is in progress.
* A decrease in pain after the injection of MSCs was observed in patients treated by radiotherapy for breast cancer, radiation burns, and radiotherapy over-dosage.
* Four patients, were treated with MSCs after receiving overdose pelvic irradiation for prostate cancer. A decrease in pain (EN score), bleeding and diarrhea was observed.

MSCs will represent a promising alternative strategy in the treatment of severe enteritis, rectitis and cystitis after radiotherapy, and may avoid surgical treatment and may diminish the adverse effect of PRD in terms of chronicity, morbidity, mortality and health costs.

DETAILED DESCRIPTION:
-Chemo-radiation enhances survival but also increases the risk of PRD. The result will be an increasing

* Cost for society (repeated hospitalization for palliative care)
* An ethical problem to help these patients with irreversible degraded quality of life.

Results from conventional therapies for PRD reveal a poor long-term efficacy:

i. Coagulation by plasma argon is insufficient, 58% at 6 months; ii. The efficacy of formalin is questionable (48%), as is 5-amino-salicylate, sulfasalazine, vitamin E and pentoxifylline ; iii. The efficacy of short chain fatty acids and hyperbaric oxygen therapy is low (40%); iv. Steroids are of limited efficacy (37%). v. A surgical operation in an irradiated field is associated with difficult or impossible healing as well as with risks of infection (mortality of 5% within 40 months) Furthermore, conventional therapies are palliative and badly tolerated. More effective approaches are thus crucial.

* PRD unfortunately remains a major side effect of radiotherapy and there is no established effective treatment. Consequently, the recruitment of the aforementioned number of patients by participating radiotherapy centers is ensured.
* MSC therapy is a safe and suitable option in severe PRD.

  * The investigators propose a proof of concept.
  * MSC production and injection protocol has already been successfully employed in compassionate therapy on four patients, who suffered from chronic and fistulizing colitis, after radiotherapy for prostate cancer.
* PRISME is a network project which includes St Antoine Hospital, INSERM (National Institute of Health and Medical Research), EFS (French Blood Establishment ), CTSA (Army Centre of Blood Transfusion) ECellFrance, IRSN (Institute for Radiological Protection and Nuclear Safety), IGR (Gustave Roussy Institute), and Institute of cancerology of west France. Our consortium has robust experience of the treatment of radiation damages, preclinical models and the medical management of PRD using biotherapy. Clinical and scientific achievements, previous collaborations of the different groups and preliminary partner's data assure the fulfillment of the program.

  * Patient selection will be performed by the six radiotherapy centers participating in this study. The expected recruitment per center had been concluded from the average number of potentially eligible patients treated and surveyed in each of the following centers (St Antoine Hospital, Gustave Roussy Institute, Institute of cancerology of west France).
  * The ECellFrance platform will ensure MSC production. This platform includes two locations in Parisian region: EFS (in the city of Creteil) and CTSA.
  * Support, trials and intervention protocols will be handled in the Department of Clinical Hematology at St Antoine Hospital, renowned for its expertise in the treatment of overdosed radiation therapy patients, i.e. Epinal cases) and which has managed a PHRC using MSCs.
  * Participation of a research group with robust experience in stem cells, transplantation (Research centre Saint Antoine, INSERM) and radiobiology, cell therapy treatment of radiation accidents (IRSN, CTSA). These groups will carry out the characterization of the biological activity and immunological properties of the native MSC bone marrow tissue in vitro (INSERM) and in vivo (IRSN) and immunological monitoring of patients treated with the MSC (INSERM).

It is expected to achieve the healing of chronic refractory diseases, leading to lower health expenses by reducing patient treatment and hospitalization, and to an increase in their quality of life by a:

* Decrease in rectorrhagia and hematuria, pain, drug-consumption;
* Inhibition of hemorrhagic syndromes and chronic inflammation accompanied by a sustained fistulization arrest due to the repairing capability of MSC.

The expected results for the public will be the healing of chronic refractory diseases, leading to lower health expenses by reducing patient treatment and hospitalization, and to an increase in their quality of life.

Hypothesis: MSC injections provide an efficient alternative approach in the treatment of PRD for patient refractories to conventional treatments.

Patient study scheduled:

D-60: Screening by 6 radiotherapy centers. D-1: Inclusion in Saint Antoine Hospital. D0, D7 and D14: IV MSC injection (2x106 - 6x106/kg MSC). M2 and M4: follow-up visit. End of patient's participation to the study at M4. Total number of scheduled patients: 12 patients suffering from PRD. Simon minimax plan, P0=25%, P1=60%, Alpha=5% and Beta=20%.

Stopping rules:

Step 1: (n1=5) inclusion of 5 patients r1=1: if the number of success is <2, the study will end for MSC inefficacy. If the number of success is ≥2, proceed to step 2. Step 2: (n2=7) inclusion of up to 7 patients r2=5: as soon as the number of successes reaches 6 (>r2), inclusions will be discontinued and MSC will be considered as sufficiently promising for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and <80 years;
* Any pelvic cancerous pathology irradiated with a history of pelvic complications of grade > 2 LENT SOMA scale);
* Absence of metastasis objectified by bone scintigraphy;
* After failure following at least three lines of conventional treatment;
* Good physical condition (WHO-performance status 0-1)

Exclusion Criteria:

* Pregnancies (Pregnancy test carried out during the inclusion examination).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Decrease of one grade on the LENT SOMA | 4 months after the first injection of MSCs
  Decrease of one grade for rectorrhagia or hematuria on the LENT SOMA scale (Late Effects Normal Tissue Task Force -Subjective, Objective, Management, Analytic), 4 months after the first injection of MSCs.

SECONDARY OUTCOMES:
The effect of treatment on analgesic drug consumption (analgesic, opiates). | 4 months after the first injection of MSCs
  Frequency of drug consumption (analgesic, opiate)
The effect of treatment on quality of life with SF36 questionnaire | 4 months after the first injection of MSCs
  Quality of life evaluated by SF36 questionnaire (short form survey)
The effect of treatment on quality of life with HADS questionnaire | 4 months after the first injection of MSCs
  Quality of life evaluated by questionnaire Hospital Anxiety and Depression Scale (HADS)
The effect of treatment on pain | 4 months after the first injection of MSCs
  Mean pain intensity evaluated by Visual Analogue Scale (VAS) during the week prior to the visit.
Frequency of diarrhea | 4 months after the first injection of MSCs
  diminution of the frequency of diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad MOHTY, PhD, Principal Investigator — mohamad.mohty@inserm.fr
Locations (1):
- Hématologie et thérapie cellulaire, Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided